CLINICAL TRIAL: NCT05736744
Title: Effect of Magnesium Sulphate Pretreatment on the Onset and Duration of Intense and Deep Neuromuscular Block of Rocuronium Versus Cis-Atracurium in Pediatric Abdominal Surgery
Brief Title: Effect of Magnesium Sulphate Pretreatment in Pediatric Abdominal Surgery
Acronym: MgSO4/MR
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-2022-200028
Record Dates: First submitted 2023-01-20; First posted 2023-02-21 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Muscle Relaxation
MeSH Terms: interventions — Magnesium Sulfate; cisatracurium

STUDY DESIGN:
Intervention Model Description: To compare the effect of magnesium sulphate pretreatment on the onset and duration of intense and deep neuromuscular Block of rocuronium versus Cis-Atracurium and on the period of no response to nerve stimulation in children undergoing elective laparoscopic surgeries.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The dose of the administered muscle relaxants will be given by an investigator not included in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cis/atracurium/saline placebo (Placebo Comparator): 1. The patients will receive 100 ml saline 0.9% at an infusion rate 5 ml/min-1) administered 20 min. before induction of anesthesia.
  2. cisatracurium will be administered for intubation at a dose of 0.15 mg/kg IV and Maintenance at a dose of 0.03 mg/kg IV
  Interventions: Drug: Cis-Atracurium
- Cis-Atracurium/MgSO4 (Active Comparator): 1. The patients will be pretreated with magnesium sulphate infusion (30 mg kg-1, total volume 100 ml, infusion rate 5 ml min-1) 20 min. before induction of anesthesia.
  2. Cis-Atracurium will be administered at 0.1-0.15 mg/kg IV bolus for intubation and maintenance at a dose of 0.03 mg/kg iv on fixed intervals.
  Interventions: Drug: MgSO4; Drug: Cis-Atracurium

INTERVENTIONS:
Drug: MgSO4 — The patients will be pretreated with magnesium sulphate infusion (30 mg kg-1, total volume 100 ml, infusion rate 5 ml min-1) 20 min. before induction of anesthesia.
  Other Names: Magnesium Sulfate
  Arms: Cis-Atracurium/MgSO4
Drug: Cis-Atracurium — Cis-Atracurium will be administered at 0.1-0.15 mg/kg IV bolus for intubation and maintenance at a dose of 0.03 mg/kg iv on fixed intervals.
  Other Names: Nimbex

SUMMARY:
In this study, the investigators will compare the effect of magnesium sulphate pretreatment on the onset and duration of intense and deep neuromuscular Block of rocuronium versus Cis-Atracurium and on the period of no response to nerve stimulation in children undergoing elective open abdominal surgeries.

DETAILED DESCRIPTION:
Deep neuromuscular blockade is known to improve surgical conditions in procedures such as abdominal or pelvic laparoscopic surgery, laparotomy and laryngeal surgery. In addition, deep neuromuscular blockade enables a reduction in pneumoperitoneal pressure, postoperative pain and the incidence of intra-operative and postoperative adverse events. Correspondingly, the use of deep neuromuscular blockade is increasing, and for its maintenance neuromuscular monitoring is essential; the use of neostigmine may also be helpful in achieving a rapid recovery. Magnesium sulphate has gained prominence as an adjuvant drug in multimodal anesthesia and pain medicine. It has several clinical indications, including attenuation of the adrenergic response to tracheal intubation and improved peri-operative analgesia. Magnesium sulphate also enhances the action of non-depolarizing neuromuscular blocking drugs, resulting in potentiation of neuromuscular blockade (NMB).The site of magnesium potentiation of neuromuscular blocking drugs is the motor end plate, where magnesium reduces the release of prejunctional acetylcholine, thereby decreasing the muscle membrane excitability. However, limited data exist concerning the effect of magnesium sulphate on the duration of deep or intense NMB and on the period of no response to nerve stimulation. In this study, the investigators will compare the effect of magnesium sulphate pretreatment on the onset and duration of intense and deep neuromuscular Block of rocuronium versus Cis-Atracurium and on the period of no response to nerve stimulation in children undergoing elective open abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Age group 2-12 years old
2. Both genders
3. Children who will be scheduled to undergo elective laparoscopic surgeries.
4. Patients with American Society of Anesthesiologist physical status classification of 1 or 2-

Exclusion Criteria:

1. Patients who are beyond the selected age group.
2. Patients on medications that interfered with muscle activity.
3. Allergy to medications used in this study.
4. Neuro-muscular diseases.
5. Renal or hepatic impairment.
6. Hypermagnesemia (>2.5 mmol) or hypomagnesemia (<1.7 mmol).
7. Parental refusal to participate in the study

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The time of no response to nerve stimulation (seconds) | Intraoperative
  Neuromuscular monitoring will be performed using acceleromyography with the TOF-Watch SX (Organon Ireland Ltd, Dublin, Ireland). Period of no response will be defined as the time period with no response to TOF stimulation (intense and deep NMB).

SECONDARY OUTCOMES:
Duration of deep NMB (seconds) | Intraoperative
  The time period from the reappearance of the first response to PTC stimulation to the reappearance of the first response to TOF stimulation.
The duration of moderate NMB (seconds) | Intraoperative.
  the time period from the reappearance of the first response to PTC stimulation to the reappearance of the first response to TOF stimulation one to three out of four twitches.
NMB onset time (in seconds). | Intraoperative.
  The time elapsed, in minutes, from the start of the administration of muscle relaxant; cis-atracurium or rocuronium injection to 95% of T1 depression.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Abdel-Ghaffar, MD, Principal Investigator — Professor of anesthesia and intensive care, faculty of medicine, Assiut university, Assiut, Egypt.
Locations (2):
- Egypt (2):
  - Pediatric hospital, faculty of medicine, Assiut university, Asyut, Assiut Governorate
  - Pediatric hospital, Asyut, Assiut Governorate

IPD SHARING:
Plan to Share IPD: No